CLINICAL TRIAL: NCT02658903
Title: Prevention of Catheter Associated Lower Urinary Infections Using the Oxys Indwelling Catheter
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oxys Medical AG (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Oxys-01
Record Dates: First submitted 2015-11-20; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Infections
Keywords: Foley; Infection; Hospital acquired; catheter associated; urinary
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study arm with Oxys-Cathter (Experimental): The study group is treated with a modified urinary catheter, which delivers electromagnetic therapy to prevent and treat bacterial colonization during the study period. The intervention is the insertion of the study urinary catheter (foley) into the bladder.
  Interventions: Device: Oxys Catheter
- Control-arm with commercial catheter (Other): The control group is treated with a commercial urinary catheter. The intervention is the insertion of the control urinary catheter (foley) into the bladder,
  Interventions: Device: Covidien Mona-Therm Foley catheter

INTERVENTIONS:
Device: Oxys Catheter — The study catheter is inserted over the urethra in the bladder as a foley catheter. The study foley catheter delivers electromagnetic therapy.
  Arms: Study arm with Oxys-Cathter
Device: Covidien Mona-Therm Foley catheter — The control arm catheter is inserted over the urethra in the bladder. The control catheter is a Mona-Therm catheter from Covidien.
  Arms: Control-arm with commercial catheter

SUMMARY:
The safety and efficacy of a urinary catheter designed to prevent catheter associated urinary infections is studied.

DETAILED DESCRIPTION:
This study is an open randomized controlled trial of 4 weeks duration. The intervention is a novel urinary catheter with an electromagnetic therapy to prevent catheter associated infections. The catheter is used in patients which require longterm urinary catheterization over at least 1 month.

The endpoint is bacteriological exam and the laboratory is blinded to the therapy status. Weekly urinary cultures are drawn and a sonication culture of the catheter tip is performed to detect and characterize the biofilm. A colonization rate of >95% is anticipated in the control arm. Therefore a 50% reduction in colonization can be detected with 54 patients, a 90% reduction in colonization can be detected with 20 patients with a power of 0.9.

ELIGIBILITY:
Inclusion Criteria:

* Patient with need for an indwelling urinary catheter to be placed at least for 4 weeks, which are willing and capable to provide informed consent. Most patients have spinal cord injury and are treated by the prinicpal investigator.

Exclusion Criteria:

* Need for antibiotic treatment for any infections
* Urological intervention or need for catheter change within study duration of 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial biofilm on catheter, assessed by ultrasonic culture of catheter tip removed at the end of the study. | 4 weeks

SECONDARY OUTCOMES:
Significant bacteriuria assessed by weekly bacterial cultures. | every week during 4 weeks
Clinically symptomatic catheter associated lower urinary infections. | 4 weeks
occurence of adverse events | within 4 weeks
  safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kessler, MD, Principal Investigator — Universitätsklinik Balgrist Zürich
Locations (1):
- University Hospital Balgrist, Zurich, Canton of Zurich, Switzerland